CLINICAL TRIAL: NCT05980624
Title: The Impact of Oral Nutrition Supplements on the Clinical Outcomes in Gastrointestinal Cancer Patients Undergoing Chemotherapy
Brief Title: ONS in Gastrointestinal Cancer Patients Undergoing Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, ALshaimaa Ibrahim Rabie, Clinical nutrition pharmacist, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FMBSUREC/09072023/Rabie
Record Dates: First submitted 2023-07-22; First posted 2023-08-08 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-03

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (No Intervention): nutrition counselling plus Standard chemotherapy only. Patients will undergo only standard chemotherapy for 3 months
- Group B (Experimental): nutrition counselling plus standard chemotherapy adding oral nutrition supplements as described in manufacturer label daily for 3 month and
  Interventions: Dietary Supplement: oral nutrition supplement

INTERVENTIONS:
Dietary Supplement: oral nutrition supplement — patients receive ONS 300kcal in daily basis
  Arms: Group B

SUMMARY:
The study hypothesizes that the addition of oral nutrition supplement concurrent chemotherapy treatment to the GI cancer patients will improve the prognosis of cancer cachexia, improve health state quality of life and increase chemotherapy tolerance

DETAILED DESCRIPTION:
Malnutrition is a major public health issue in low- and middle-income countries and forms part of the United Nations 2030 Agenda for Sustainable Development Goals .Cancer is a systemic disease, since even in the early stages malignancies are accompanied by homeostatic imbalance, including metabolic deregulation and increased catabolism. These abnormalities may initially seem poorly discernible in the clinic, but with disease progression they may aggravate; and may cause overt cancer-related cachexia.GI cancers show higher mortality than any other kind of cancer. In 2020, they accounted for an estimated 3.5 million deaths worldwide, with a further 5.0 million new cases diagnosed in the same year . Colorectal cancer (CRC) is the most common type of GI cancer, being the third most common of all organ cancers after lung and breast cancers, whereas gastric, liver, esophageal, and pancreatic cancers are ranked the fifth, sixth, eighth, and 12th most commonly diagnosed cancers, respectively

ELIGIBILITY:
Inclusion Criteria:

-

GI cancer patients will be included in the study if they meet the following criteria:

1. Confirmed cancer diagnosis any stage or metastatic confirmed by radiological and pathological or by clinical evaluation receiving neo/adjuvant chemotherapy treatment.
2. Age above 18 years old
3. Be accessible for chemotherapy treatment and follow-up
4. Availability to administer oral supplements
5. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2
6. Life expectancy ≥3 months.
7. Written informed consent according to the local Ethics Committee requirements
8. Willing to fill Nutrition questionnaires.
9. Negative pregnancy test for pre-menopausal women before inclusion in the trial

Exclusion Criteria:

* The patients will be excluded from the study if they have the following criteria:

  1. Known hypersensitivity reaction to the investigational compounds or incorporated substances
  2. patients who are unlikely to comply with trial requirements (eg, confusion, psychological or mood disturbances ,alcoholism)
  3. Pregnancy or lactating
  4. Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent
  5. Age < 18 years
  6. Indication to or ongoing artificial nutrition support (totally compromised spontaneous food-intake) and incapacity or unavailability to consume ONS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-01-16 (Actual)

PRIMARY OUTCOMES:
Body Composition | 3 month
  measured by DEXA OR BIA
Anthropometric measures | 3 month
  Body mass index change
Nutrition status - scored Patient-Generated Subjective Global Assessment (PG-SGA) | 3 MONTHS
  malnutrition assessment tool. ( 0-1 )No intervention required at this time. Re-assessment on routine and regular basis during treatment.
  (2-3) Patient & family education by dietitian, nurse, or other clinician with pharmacologic intervention as indicated by symptom survey and lab values as appropriate. (4-8) Requires intervention by dietitian, in conjunction with nurse or physician as indicated by symptoms .
  * 9 Indicates a critical need for improved symptom management and/or nutrient intervention options

SECONDARY OUTCOMES:
Laboratory data values mean and standard deviation | 3 months
  Albumin and CRP ,total protein
overall response rate | 6 months
  complete response or progression and regression percentage of participants
common adverse effects | 6 months
  Git toxicity , hematologic toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Alshaimaa Rabie, Principal Investigator — Beni-Suef University
Locations (1):
- Beni suef university hospital, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No